CLINICAL TRIAL: NCT00125125
Title: Efficacy and Tolerability of Fluvastatin in Adults With Dislipidemia With History of Muscle Problems Due to Other Previous Statin Intake
Brief Title: Fluvastatin in Adults With Dislipidemia With History of Muscle Problems
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXUO320B2406
Record Dates: First submitted 2005-07-28; First posted 2005-07-29 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Dyslipidemia
Keywords: Dyslipidemia, adults, fluvastatin
MeSH Terms: conditions — Dyslipidemias | interventions — Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin

SUMMARY:
The purpose of the study is to find a good therapy for patients who need to be treated for high cholesterol and who have difficulty tolerating other statins (such as pravastatin, simvastatin, lovastatin, atorvastatin, rosuvastatin) due to muscle pain.

ELIGIBILITY:
Inclusion Criteria:

* Dyslipidemia
* History of Myalgia

Exclusion Criteria:

* Previous treatment with fluvastatin
* Age < 18 years

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2005-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in low density lipoprotein cholesterol after 12 weeks

SECONDARY OUTCOMES:
Tolerability as assessed by muscle-related adverse events, and muscle-related adverse events leading to discontinuation
Change from baseline in total cholesterol, triglycerides, high density lipoprotein cholesterol, and lipoprotein subtypes after 12 weeks
Number of patients who reach target LDL after 12 weeks
Change from baseline in marker of inflammation after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (2):
- Novartis, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Derived] Stein EA, Ballantyne CM, Windler E, Sirnes PA, Sussekov A, Yigit Z, Seper C, Gimpelewicz CR. Efficacy and tolerability of fluvastatin XL 80 mg alone, ezetimibe alone, and the combination of fluvastatin XL 80 mg with ezetimibe in patients with a history of muscle-related side effects with other statins. Am J Cardiol. 2008 Feb 15;101(4):490-6. doi: 10.1016/j.amjcard.2007.09.099. Epub 2007 Dec 20. PMID 18312764